CLINICAL TRIAL: NCT05656417
Title: Individual Variability of Experimental Gingivitis Response: a Parallel-group Cohort Study
Brief Title: Individual Variability of Experimental Gingivitis Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Unilever R&D (Industry); Guy's and St Thomas' NHS Foundation Trust (Other); Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Sponsor
Other Study IDs: 316902
Record Dates: First submitted 2022-11-25; First posted 2022-12-19 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-03

CONDITIONS: Gingivitis; Oral Disease
Keywords: Experimental gingivitis; Periodontal disease; Gingival disease; Infectogenomics; Oral health; Dental plaque
MeSH Terms: conditions — Gingivitis; Mouth Diseases; Periodontal Diseases; Gingival Diseases; Dental Plaque

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will include saliva, whole blood, serum, sub- and supra- gingival plaque, gingival crevicular fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Haplotype 1: Participants will attend a screening visit where they will provide a saliva sample for DNA sequencing. Participants will then be separated into two groups based on their gene profile. Participants in Group 1 will have a specific haplotype of the gene of interest. The groups will undergo a 2-week period of thorough oral hygiene and prophylactic treatment to achieve excellent gingival health. Participants in both groups will then cease all oral hygiene for a period of 3 weeks, where a state of gingivitis will develop. At the end of the 3 weeks, normal oral hygiene will be reinstated and prophylactic treatment offered as required for a further 2 weeks.
  Interventions: Behavioral: Temporary cessation of all oral hygiene
- Haplotype 2: Participants will attend a screening visit where they will provide a saliva sample for DNA sequencing. Participants will then be separated into two groups based on their gene profile. Group 2 will comprise of participants who possess a second distinct haplotype in the same gene of interest as Group 1. This group will undergo the same study procedures as Haplotype Group 1.
  Interventions: Behavioral: Temporary cessation of all oral hygiene

INTERVENTIONS:
Behavioral: Temporary cessation of all oral hygiene — Participants will refrain from all oral hygiene for 3 weeks.
  Other Names: Experimental gingivitis

SUMMARY:
The study aims to investigate the genetic cause of the variability between individuals seen in the development of the gum disease, gingivitis. This will be carried out through a 3 week programme where all oral hygiene is ceased, allowing 'experimental gingivitis' to develop, followed by a period of recovery when tooth cleaning is restored. Clinical assessments and biological samples will be taken during the course of the study for further analysis.

DETAILED DESCRIPTION:
The purpose of the project is to investigate the factors which influence the oral disease, gingivitis. Gingivitis is the inflammation (swelling, redness, pain) of the gums, caused by the build-up of bacteria in the mouth. Research shows that the severity, extent and rate of development of gingivitis varies considerably between individuals. The aim of this project therefore is to investigate if an individual's DNA contributes to this range in outcomes and what impact it has on the human and bacterial cells in the mouth. This will be investigated through a period where all tooth brushing and oral hygiene will cease, and the changes in the mouth measured as the temporary 'experimental gingivitis' develops. Clinical measurements will include plaque build-up, levels of inflammation and bleeding scores, while samples of blood, saliva and plaque will be used to quantify changes in inflammatory markers and bacterial community composition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35
* Caucasian
* No history of periodontitis/periodontal treatment (based on self-reported history)
* Medical history clear of cardiovascular disease, diabetes, cerebrovascular disease, kidney or liver disease, cancer, HIV, Tuberculosis and Hepatitis C (self-reported)
* Never smoker, e-cigarettes or nicotine gum use (self-reported). Individuals who rarely socially smoked more than 5 years ago would be permitted to participate.
* Minimum of 24 teeth present
* Be willing and competent (verbally and cognitively) to give written informed consent and complete a medical history form
* Be willing and physically able to carry out all study procedures
* Not have had a scale and prophylaxis in the previous month or have one scheduled prior to the end of the study
* Participant in good periodontal health, based on:

  1. absence of interproximal probing pocket depths (PPD) and clinical attachment level (CAL) > 3mm (with the exception of distal surfaces of third molars in the presence of impacted third molars) at the screening visit.
  2. bleeding on probing (BOP) < 30% at the Screening visit and BOP <10% at Day -7.

Exclusion Criteria:

* Currently taking part in other clinical trials
* Pregnant or breastfeeding women
* Taking medications including systemic anti-inflammatory medication within 3 months of the study (NSAIDs, no more than once per week and not in the week before sample collection, is permitted)
* Systemic antibiotic intake within 6 months
* Psychiatric conditions affecting participation in the study
* The participant is also a member of staff who is part of the study team
* Current orthodontic treatment
* Regular consumption of alcohol exceeding the government recommended levels
* Denture wearer/presence of dental implants/bridges
* Have oral piercings
* Obvious signs of untreated caries
* Taking dietary supplements (e.g. multivitamins; antioxidants; fish oils)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Gingivally healthy young adults
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Löe-Silness Gingival Index: Min 0 - Max 3; Higher score indicates more gingival inflammation and a worse outcome. | Intervals over 6 weeks.
  Change from baseline.

SECONDARY OUTCOMES:
Silness-Löe Plaque Index: Min 0 - Max 3; Higher score indicates more plaque accumulation and a worse outcome. | Intervals over 6 weeks.
  Change from baseline.
Bleeding on Probing: Min 0 - Max 1; Higher score indicates bleeding at the gingival site and a worse outcome. | Intervals over 6 weeks.
  Change from baseline.
Microbial dysbiosis (detection and counts of subgingival microbes). | Intervals over 6 weeks.
  Change from baseline.
Inflammatory markers (e.g. matrix metalloproteinase-8 and IL-1β) in blood, gingival crevicular fluid and saliva samples: Higher levels indicate a greater degree of gingival inflammation. | Intervals over 6 weeks.
  Change from baseline. Measured by enzyme-linked immunosorbent assay (units: ng/mL) in each sample type.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Nibali, PhD, Principal Investigator — King's College London
Locations (1):
- Centre for Host-Microbiome Interactions, Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
A data sharing agreement is in place with a funder of the project, Unilever plc. Anonymised participant demographics will be linked to the data, such as year of birth and sex.